CLINICAL TRIAL: NCT03548181
Title: Feasibility & Effect of a Tele-rehabilitation Program in Idiopathic Pulmonary Fibrosis (IPF)
Acronym: 3-IPF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Eurostars (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3-TELE IPF
Record Dates: First submitted 2018-05-24; First posted 2018-06-07 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-05

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Tele-rehabilitation
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: The study is a prospective, randomized controlled trial comparing the effects of tele-rehabilitation and standard treatment in patients with IPF
Who Masked: Participant, Outcomes Assessor
Masking Description: The study is a randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group "tele-rehabilitation" (Experimental): Each patient will have the opportunity to have minimum one Video Consultation (VC) per week the first month, one VC each second week the second month one VC a month the rest of the trial.
  Workout Sessions with a Virtual Physiotherapist Agent (VPA): The patient will train according to what is decided by the physiotherapist and the patient in the VC or chat meetings. Normally, the patients will train 10-20 minutes daily at home with its individual and tailored VPA. Instead of ergometer bike training, the patient will receive some easy training tools such as elastics, weights and a fitness-step that can be used in the different exercises showed by the VPA to reach the same intensity of workout. The VPA will then be animated to motivate and encourage the patient to exercises at home. A digital diary will automatically register the data obtained by the system on patient's performance.
  Interventions: Behavioral: Virtual Autonomous Physiotherapist Agent (VAPA)
- Control (Active Comparator): Patients will be followed, but they do not get any other kind of treatment comparable to the intervention group treatment.
  Interventions: Behavioral: Virtual Autonomous Physiotherapist Agent (VAPA)

INTERVENTIONS:
Behavioral: Virtual Autonomous Physiotherapist Agent (VAPA) — A Virtual Autonomous Physiotherapist Agent is going to gide and motivate the patient to train physically at home.
  Other Names: VAPA

SUMMARY:
Introduction Idiopathic Pulmonary Fibrosis (IPF) is a progressive fibrotic lung disease of unknown cause with a median survival of 3-5 years. As the disease progresses, worsening of lung function and gas exchange impairment cause hypoxemia during physical activity leading to a downward spiral; dyspnea and fatigue lead to a reduction in daily physical activities, exercise tolerance, muscle strength and quality of life. Problems reported by IPF patients are social isolation, increased level of dependency and immobility.

There is no curative treatment for IPF, but pulmonary rehabilitation (PR) is recommended by expert opinion for the majority of IPF patients in order to improve quality of life and exercise tolerance. There are, however, no official PR programs for IPF patients and they therefore either participate in PR programs patients with chronic obstructive lung diseases (COPD) or train by themselves in fitness centers without guidance. PR for COPD is mostly offered in specialized clinics with an average duration of 8 weeks. Not all patients with IPF are fit for these programs or want to participate in an extensive external program due to, among other reasons, distance to the clinic. Tele-rehabilitation may offer these patients an alternative.

New technologies in healthcare that can treat patients from a distance are implemented in these years. Tele-rehabilitation has been shown to be feasible in patients with lymphedema, COPD, orthopedic diseases (lower back, knee and shoulder). To ensure that all IPF patients are offered the possibility to participate in IPF specific rehabilitation programs, even though they live far away from expert ILD centers, tele-rehabilitation might be an alternative to participation in COPD rehabilitation programs. There have so far been no studies on the feasibility effect of tele-rehabilitation in IPF.

Aim To assess the feasibility and effect of tele-rehabilitation with a new and innovative TR platform (NITRP) compared to standard treatment with respect to exercise capacity, quality of life and activities of daily living in patients with IPF.

Method & material The study is a prospective randomized controlled trial comparing the effects of tele-rehabilitation and standard treatment in patients with IPF. 24 patients with IPF will be randomized in two groups, and the intervention group trained by tele-rehabilitation for 12 weeks with follow-up after training at 3 and 6 months. The control group will follow the usual control program for IPF patients that only involves outpatient visits approximately every 3rd month. The intervention group will recieve tele-rehabilitation.in the form of video consultations- and chat sessions with a real physiotherapist and workout sessions with a virtual physiotherapist agent. They will also train with virtual reality glasses or tablets that show the actual exercises in the training program.

Patients will be tested with pulmonary function parameters, 6 minute walk test, a pedometer registering steps walked in 7 days, King's brief ILD questionnaire (a disease specific quality of life questionnaire), the General Anxiety Disorder Score (GAD-7) (measures the presence and severity of general anxiety disorder) and the SGRQ-IPF, a disease specific, self-administered questionnaire for IPF, all at baseline, after 12 weeks of intervention, 3 and 6 months after cessation of the program

DETAILED DESCRIPTION:
Background:

Idiopathic Pulmonary Fibrosis (IPF) is a progressive fibrotic lung disease of unknown cause with a median survival of 3-5 years (Raghu et al. 2011). As the disease progresses, worsening of lung function and gas exchange impairment cause hypoxemia during physical activity leading to a downward spiral; dyspnea and fatigue lead to a reduction in daily physical activities, exercise tolerance, muscle strength and quality of life (Behr et al. 2013)(Holl and Hill, 2008). Problems reported by IPF patients are social isolation, increased level of dependency and immobility (Bajwah et al. 2012)(De Vries et al. 2001).

No curative treatment exists (Raghu et al. 2011). Pulmonary rehabilitation (PR) is recommended by expert opinion for the majority of IPF patients to improve quality of life and exercise tolerance (Raghu et al. 2011) (Behr et al. 2013). These programs are mostly offered in specialized clinics with an average duration of 8 weeks (Holl et al. 2008)(Nishiyama et al. 2008)(Jastrzebski et al. 2006)(Huppmann et al. 2012)(Verma et al. 2011)(J J Swigris et al. 2005). Not all patients with IPF are fit for these programs or want to participate in an extensive external program due to, among other reasons, distance to the clinic. Tele-rehabilitation may offer these patients an alternative.

Tele-rehabilitation seems to be a good approach to reach patients in low inhabited areas (Hill and Sppath, 2010), going from health care to self-care (Haarder 2011), empowering patient's awareness of their disease and increasing the flexibility patients need to acquire healthier behaviors. Tele-rehabilitation has previously been shown to be feasible in patients with lymphedema (Galiano-Castillo et al. 2014), COPD (Paneroni et al. 2014)(Tousignant et al. 2012)(Dinesen, Seeman, and Gustafsson, 2011)(Dinesen, Huniche, and Toft, 2013) and orthopedic diseases, lower back (Palacín-Marín, Esteban-Moreno, Olea, Herrera-Viedma, and Arroyo-Morales, 2013), knee (Cabana et al. 2010) (Tousignant, Moffet, et al. 2011) (Tousignant, Boissy, et al. 2011) and shoulder (Eriksson, Lindström, Gard, and Lysholm, 2009)(Eriksson, Lindström, and Ekenberg, 2011).

Tele-rehabilitation with COPD patients at home is feasible and well accepted by the patients, although technology has been perceived as difficult (Paneroni et al., 2014)(Tousignant et al.,2012). Tele-rehabilitation seems to improve the functional level as assessed by walking capacity, dyspnea, quality of life and daily physical activity (Paneroni et al. 2014). The interaction between the COPD patients at home and the healthcare professionals at the clinic through tele-rehabilitation has evolved as a dialogue channel forming a basis for mutual learning processes and new relationships (Dinesen, ersen, Hejlesen, & Toft, 2011). Preliminary evaluations from tele-rehabilitation initiatives in Scotland showed tele-rehabilitation to be more cost effective with patients living in remote areas than with the outreach- or centralized model (Hill and Sppath, 2010).

Thus, in order to ensure that all IPF patients are offered the possibility to participate in IPF specific rehabilitation programs even though they live far away from expert centers, tele-rehabilitation might be an alternative to standard rehabilitation programs or to, as often happens, participation in COPD rehabilitation programs. There have so far been no studies on the feasibility effect of tele-rehabilitation in IPF.

Hypothesis Tele-rehabilitation in patients with IPF is feasible and improves exercise capacity, quality of life and activities of daily living.

Aim To assess the feasibility and effect of tele-rehabilitation with a tele-rehabilitation platform (NITRP) compared to standard treatment with respect to exercise capacity, quality of life and activities of daily living in patients with IPF.

Design:

The study is a prospective, randomized controlled trial comparing the effects of tele-rehabilitation and standard treatment in patients with IPF

Patients 24 patients with IPF followed in the outpatient clinic at the Danish Centre for Interstitial Lung Diseases at the Department of Respiratory Diseases & Allergy, Aarhus University Hospital will be recruited and randomized to participate in the study.

Inclusion criteria

In order to be eligible to participate in this study, the patient must meet all of the following criteria:

Diagnosis of either definite or possible IPF according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria Signed informed consent DLCO ≥ 30% predicted and FVC ≥ 50% predicted 6 minute walking test ≥ 150 m Adults ≥ 18 years Being clinically stable Absolute decline in DLCO & FVC should be less than 10% in the past 6 months.

Exclusion criteria

A potential patient who meets any of the following criteria will be excluded from participation in this study if:

Participation in an official rehabilitation program < 4 months before start of the study Musculoskeletal disorders Severe cardiac diseases (ejection fraction < 30%, daily angina, or otherwise specified by treating cardiologist) Unable to understand informed consent Other conditions that hamper the use of tele-rehabilitation Non-Danish speaking. Unwillingness to implement the protocol

Sample size calculation There have been no studies of tele-rehabilitation in IPF and previous studies have used other indices for evaluation of quality of life measures. Therefore, there are no data available for sample size calculation. This study will be a pilot study to estimate the effect of a tele-rehabilitation in which we aim to include 24 patients, 12 in each group

Treatment of subjects No changes in regular treatment will be done because of participating in the tele-rehabilitation study.

Investigational treatment The intervention is the use of a tele-rehabilitation program during 12 weeks. The patient's training time will be registered automatically. The control group will receive standard treatment only.

Escape medication In case of exacerbation of IPF or a respiratory tract infection, the patient will be treated to the discretion of the clinician in charge and excluded from the study. However, the patients will be offered to be included again at the moment clinical stability is reached and the patient again fulfils inclusion criteria.

Method

Randomisation, blinding & treatment allocation Randomisation will allocate patients to either the intervention or control group and will be performed electronically. The questionnaires on quality-of-life are self-administered questionnaires. Participants will be asked to complete them before talking to the physician.

Study procedures The trial will be registered in the public database of Clinical Trials.gov. All consecutive clinical stable patients with definite or possible IPF from the outpatient clinic at the Danish Center of Interstitial Lung Diseases, at the Department of Respiratory Diseases and Allergy, Aarhus University Hospital that might be eligible will be informed about the study by their respiratory physician or nurse. The patients will be asked if they are interested in participating in this study, and if so, they will receive verbal and written information. In this information the study is explained in detail. The patients have to give their informed signed consent to the principal investigator or his designee before the patient can enter the trial. After informed consent the patients will be screened during the baseline visit and physical examination, pulmonary function tests and 6 minute walk test will be performed. If pulmonary function test and 6MWT have been assessed less than 3 months or 1 month respectively, prior to the screening visit, these results can be used. Clinical stability will be assessed by the physician. If patients are eligible they will be randomized to the intervention group or control group.

At baseline all patients will be asked to complete the questionnaires on health-related quality of life and anxiety. Patients will be asked to wear a pedometer and record steps during 7 days and will be instructed not to change their daily routine while wearing this device. After returning back the pedometer patients allocated to the intervention group will receive instructions in the tele-rehabilitation program. The training program will last 12 weeks. In week 12 both groups will receive a pedometer to register steps for 7 days during the intervention. After 12 weeks, when the intervention program has ended, pulmonary function tests, 6 minute walk test and the questionnaires will be repeated.

Patients allocated to the control group will follow the same procedure except for not using tele-rehabilitation.

Patients who desaturate < 88% during the 6 minute walk test at baseline will be offered supplemental oxygen during exercise.

Follow-up 3 and 6 months after end of training will include the same parameters as at baseline: pulmonary function tests, 6 minute walk test and quality of life questionnaires.

The intervention group will undergo tele-rehabilitation as described below. After the intervention period, patients in the intervention group are invited to keep the training tools and use them as much they want with no involvement from the physiotherapist at all.

Intervention Group: Virtual Rehabilitation

The intervention group with IPF patients will follow this procedure Video Consultation (VC) Sessions: Each patient will have the opportunity to have minimum one VC per week the first month, one VC each second week the second month one VC a month the rest of the trial. Here the physiotherapist, via history will extract the information needed to calibrate the daily TR program according to the patient's physical status and needs.

Retraining breath: Patients will also be instructed to use different techniques to breath during the video consultations with the physiotherapist. The difference between the techniques used by patients with IPF and COPD is as follows: In both cases, the patient receives advice on how to the use breathing retraining techniques such as pursed lip breathing (PLB). Because COPD patients suffer from obstructed airways, the goal for them using PLB will be to increase their positive expiratory pressure (Anne E Holl, Hill, Jones, McDonald, 2012). IPF patients will be advised to use PLB with the goal of improving their breathing control and diaphragmatic effort since they do not suffer from obstructed airways and with the intention to prevent tachypnea and anxiety and to improve gas exchange (Jeffrey J. Swigris, Brown, Make, Wamboldt, 2008).

Chat Sessions: Each patient has the opportunity to chat with the physiotherapist any time via the chat module of the system. The patient and physiotherapist will be reminded via mail, anytime someone is writing in the chat, allowing the users to interact when needed.

Workout Sessions with a Virtual Physiotherapist Agent (VPA): The patient will train according to what is decided by the physiotherapist and the patient in the VC or chat meetings. Normally, the patients will train 10-20 minutes daily at home with its individual and tailored VPA. Instead of ergometer bike training, the patient will receive some easy training tools such as elastics, weights and a fitness-step that can be used in the different exercises showed by the VPA to reach the same intensity of workout. The VPA will then be animated to motivate and encourage the patient to exercises at home. A digital diary will automatically register the data obtained by the system on patient's performance.

Patients' security: In order to minimize the risks of possible accidents while performing the exercises, the patient will answer questions before and after each exercise performance that the physiotherapist can follow in real time via scales and use to calibrate the performance of the virtual physiotherapist. The patient has the opportunity to chat with the physiotherapist 24 hours per day any time if needed and for consultation reasons.

Study parameters/endpoints

Primary endpoint:

Change in the distance walked at a 6MWT measured at week 12.

Secondary endpoint:

Change in the distance walked at a 6MWT measured 3 and 6 months after cessation of the tele-rehabilitation program compared to baseline.

Change in total score in health-related quality of life measured by SGRQ-IPF at week 12, and 3 and 6 months after cessation of the tele-rehabilitation program compared to baseline.

Change in total score in health-related quality of life measured by KBILD at week 12, and 3 and 6 months after cessation of the tele-rehabilitation program compared to baseline.

Change in total score of anxiety measured by GAD-7 at week 12, and 3 and 6 months after cessation of the tele-rehabilitation program compared to baseline.

Change in component scores (symptoms, activity & impact) in health-related quality of life measured by SGRQ-IPF at week 12, and 3 and 6 months after cessation of the tele-rehabilitation program compared to baseline.

Change in the number of steps walked measured by a pedometer. Cost of the tele-rehabilitation program

End-point parameters

Pulmonary function tests (PFT):

PFT are performed as part of the routine medical follow up. The following pulmonary function indices will be registered:

Forced expiratory volume in 1 second (FEV1) Forced vital capacity (FVC) Diffusion capacity for carbon monoxide (DLCO) If DLCO cannot be measured because of cough, or other reasons, FVC should be >50% and there should be no history of known pulmonary hypertension in order to include the patient in the study. PFT are performed to prove disease stability.

Screening will be planned at the day of the routine visit. PFT form this day or performed within 3 months of this visit will be used. At 12 weeks, PFT will be repeated to check clinical stability. These PFT can replace the usual routine medical follow-up which is normally scheduled at 12 weeks intervals at our clinic.

6 minute walk test: Data of 6 minute walk test (6MWT) will be collected at screening or results of a test < 1 months prior to baseline. 6MWT will also be performed after 12 weeks and after 3 and 6 months after cessation of the program to assess exercise performance.

Pedometer:

To assess the physical activity status of the patient, measurement of the number of steps walked is an indication of the magnitude of physical activity. In controlled laboratory settings, the Yamax Digi-walker SW-200 has consistently been shown to be among the most accurate. It's a small device worn on the belt or waist and responds to vertical accelerations of the hip during gait cycles.

Questionnaires:

At baseline, and after 12 weeks and 3 and 6 months, the patient will be asked to self-administer the following questionnaires on quality of life and general well-being:

K-BILD The King's Brief Interstitial Lung disease health status questionnaire is a disease specific, validated, self-completed health status questionnaire that is comprised of 15 items. It has three domains: psychological, breathlessness, activities and chest symptoms. The KBILD domain and total score ranges are 0-100; 100 = best. Appendix 1.

SGRQ-I The SGRQ-I is a disease specific, self-administered questionnaire with 50 items comprising three domains, symptoms, activity impacts, each scored from 0-100, with higher scores corresponding to worse health related quality of life. Originally designed for patients with obstructive disease, the SGRQ-I has been developed for IPF patients and found to be a valid measure of health related quality of life. Appendix 2.

GAD-7:

The General Anxiety Disorder Score measures the presence and severity of general anxiety disorder. It is a 7 self-rated items, each item scores 0-3 (not at all, several days, more than half the days, nearly every day); total score range 0-21 (appendix 3).

IPF exacerbations:

The number of exacerbations and visits to the general practitioner, emergency room or hospital during rehabilitation and follow-up will be registered, first via a diary and corroborated then by short interviews performed during follow up at 12 weeks, and after 3 and 6 months after cessation of training.

Cost:

The average cost of the hospital rehabilitation program and transportation per patients for an eight weeks standard and tele-rehabilitation program and transportation will be calculated.

Statistical analysis The data will be analyzed according to the intention-to-treat principle and per-protocol.

Ethical considerations Regulation statement The study will be conducted according to the principles of the Declaration of Helsinki (59th WMA General Assembly, Seoul, Korea, October 2008) and in accordance with the Medical Research Involving Human Subjects Act (WMO). The trial has been reported to and approved by the Data Protection Agency in Denmark.

Recruitment and consent All IPF patients in a follow-up program at the Department of Respiratory Diseases and Allergy, Aarhus University Hospital that might be eligible will be informed about the study by their respiratory physician or nurse when evaluated at a scheduled follow-up visit. The patients will be asked if they are interested in participating in this study, and if so, they will receive verbal and written information. An enrolment letter will also be hung up at the outpatient clinic to inform potential participants about the project. The study is explained in detail in the patient information. Potential participants are entitled to at least one day of consideration time before they decide whether to participate in the trial. They have the right to be accompanied by a family member, friend or acquaintance for the oral information they will receive previous to the enrolment. The patients have to give their informed signed consent to the principal investigator or his designee before the patient can enter the trial..

Benefits and risks assessment, group relatedness Patients with IPF allocated to the intervention group might gain personal benefit from participating in this study because of the use of tele-rehabilitation. The potential effect of this study might affect future care of IPF patients and could lead to an improvement of quality of life by the reduction of social isolation, dependency and immobility, and to improved exercise performance. This study involves minimal risk for the subject. Previous rehabilitation studies have had no safety issues related to rehabilitation of patients with IPF of the same age and lung function impairment.

Handling and storage of data and documents All data will be held confidentially and will only be identifiable by number and not by name. Only the investigators have insight in the original patient linked to the data. The data will be stored at the Department of Respiratory Medicine and Allergy at Aarhus University Hospital. Study data will be accessible for authorized personnel only.

Publication:

Authorship must meet the Vancouver rules in which everyone who has contributed under this framework, will be named in the author list and included in the research protocol. The results will be published in international peer-reviewed journals and presented at relevant conferences. Moreover, the results will be published in other relevant media. All positive, negative and inconclusive results will be published Passed on information from the patient journal system Patient data will be passed on from the electronic patient files to the project.

Gender, age and marital status, will be passed on at the beginning of the study to compare the data at the end of the trial.

Telephone number, address and or E-mail from participants in the focus group will be passed on with the goal to contact the participant in the case there is a break in the connection via the tele rehab devices or if we need to send a new updated devices.

Health status, number of exacerbations in the last period, days of hospitalization, number of visits to the hospital or number of visits from healthcare suppliers to participants at home will be used to calculate the health care expenditure for each participant.

Economy MD, Ph.D. Elisabeth Bendstrup, MD Anders Løkke, MD, Ph.D., DMSc. consultant Ole Hilberg and physiotherapist José Cerdan has initiated this project and sought various foundations to execute this study.

Elisabeth Bendstrup, Anders Løkke and Ole Hilberg are the responsibles of the investigation for this study and have no financial ties to the donors.

The study is predominantly financed by EURO STARS Foundation (1,500,000 kr.) and Aarhus University (about 450,000 kr.).

Physio R and D, Laster Technologies, Cortrium and bookBeo are providing the technology, network, hardware, software and support needed for free.

Aarhus University Hospital provides locations and resources as needed and pays for the costs of the control group training. Aarhus University Hospital is also responsible for the administration and disbursement of funding.

Enrolled participants do not receive honorees for participating in this study. Transport costs associated with the trial will be covered by Aarhus University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study, the patient must meet all of the following criteria:

Diagnosis of either definite or possible IPF according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria Signed informed consent DLCO ≥ 30% predicted and FVC ≥ 50% predicted 6 minute walking test ≥ 150 m Adults ≥ 18 years Being clinically stable Absolute decline in DLCO & FVC should be less than 10% in the past 6 months.

Exclusion Criteria:

* A potential patient who meets any of the following criteria will be excluded from participation in this study if:

Participation in an official rehabilitation program < 4 months before start of the study Musculoskeletal disorders Severe cardiac diseases (ejection fraction < 30%, daily angina, or otherwise specified by treating cardiologist) Unable to understand informed consent Other conditions that hamper the use of tele-rehabilitation Non-Danish speaking. Unwillingness to implement the protocol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-05-30 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in the distance walked at a 6MWT measured at week 12 | 12 weeks
  Change in the distance walked at a 6MWT measured at week 12

SECONDARY OUTCOMES:
Change in the distance walked at a 6MWT | measured 3 and 6 months after cessation of the tele-rehabilitation program compared to baseline
  Change in the distance walked at a 6MWT measured 3 and 6 months after cessation of the tele-rehabilitation program compared to baseline.
Change in total score in health-related quality of life measured by SGRQ-IPF | at week 12, and 3 and 6 months after cessation of the tele-rehabilitation program compared to baseline.
  Change in total score in health-related quality of life measured by SGRQ-IPF at week 12, and 3 and 6 months after cessation of the tele-rehabilitation program compared to baseline.
Change in total score in health-related quality of life measured by KBILD | at week 12, and 3 and 6 months after cessation of the tele-rehabilitation program compared to baseline.
  Change in total score in health-related quality of life measured by KBILD at week 12, and 3 and 6 months after cessation of the tele-rehabilitation program compared to baseline.
Change in total score of anxiety measured by GAD-7 | at week 12, and 3 and 6 months after cessation of the tele-rehabilitation program compared to baseline.
  Change in total score of anxiety measured by GAD-7 at week 12, and 3 and 6 months after cessation of the tele-rehabilitation program compared to baseline.
Change in component scores (symptoms, activity & impact) in health-related quality of life measured by SGRQ-IPF | at week 12, and 3 and 6 months after cessation of the tele-rehabilitation program compared to baseline.
  Change in component scores (symptoms, activity & impact) in health-related quality of life measured by SGRQ-IPF at week 12, and 3 and 6 months after cessation of the tele-rehabilitation program compared to baseline.
Change in the number of steps walked measured by a pedometer. | at week 12, and 3 and 6 months after cessation of the tele-rehabilitation program compared to baseline.
  Change in the number of steps walked measured by a pedometer.
Cost of the tele-rehabilitation program | At week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Jose Cerdan, Aarhus, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633